CLINICAL TRIAL: NCT02269397
Title: Proof of Principle for a Diagnostic Blood Test of Recurrent Seizures
Status: Completed | Type: Observational
Sponsor: Cognizance Biomarkers, LLC (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 817914
Record Dates: First submitted 2013-07-09; First posted 2014-10-21 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Epilepsy
Keywords: Epilepsy; Seizures; Diagnosis; Diagnostic; Inflammation
MeSH Terms: conditions — Epilepsy; Seizures; Disease; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Subjects will be asked to give blood for evaluation of a diagnostic blood test for epilepsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Individuals with suspected epilepsy: The study will enroll individuals who are attending their first visit at the University of Pennsylvania for suspected epilepsy.

SUMMARY:
The primary goal of this observational study is to establish the accuracy of CNS-specific Assay for Recurrent Paroxysmal Events (CARPE) as a diagnostic blood test for epilepsy. The target population is patients who have been newly referred to the Penn Epilepsy Center or patients who are admitted to HUP for continuous video EEG monitoring. (Subjects without an epilepsy diagnosis will be included.) Subjects will be asked to provide consent, agree to allow the study team to collect information from their medical record, and to provide at least one blood sample.

ELIGIBILITY:
Inclusion Criteria:

* Male/female patients aged 12 and older
* Evaluation in at least one of the following settings:
* Newly referred to the University of Pennsylvania Penn Epilepsy Center. These patients may not have completed any diagnostic evaluation at Penn, other than an initial physician consultation, prior to enrollment and must agree to allow the study team to collect records regarding their diagnostic evaluations (including EEG). Diagnostic evaluations may take place at Penn or outside sites
* All patients who are admitted to the University of Pennsylvania for continuous video EEG (cVEEG) monitoring

Exclusion Criteria:

* Patients who, in the opinion of the investigator or the patients neurologist, are unable to give Informed Consent due to mental impairment or any other reason AND do not have a LAR who can give Informed Consent on their behalf. Patients aged 12-17 (inclusive) must provide assent if they are mentally capable of doing so, and must also have a caregiver who provides Informed Consent on their behalf
* Patients who, in the opinion of their neurologist at the University of Pennsylvania, are not good candidates for donating blood for any reason

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects aged 12 years and older who are attending their first visit to the University of Pennsylvania's Epilepsy Center for diagnostic purposes
Sampling Method: Non-Probability Sample
Enrollment: 371 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2015-07-14 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
Epilepsy diagnosis (CARPE) blood test for determining the presence of epilepsy ad in doing so, determine the threshold for diagnosis | 2 years
  Epilepsy diagnosis determined by three epileptologist's review of subject's medical records

CONTACTS AND LOCATIONS:
Overall Officials: Peter Crino, MD, PhD, Study Director — Cognizance Biomarkers, LLC
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

DOCUMENTS (2):
  • Informed Consent Form (2015-04-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT02269397/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2014-10-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT02269397/Prot_SAP_001.pdf